CLINICAL TRIAL: NCT05563987
Title: The Effects of an Acceptance-based Diabetes Education (ACT-DE) Programme for Adults With Type 2 Diabetes on Diabetes Distress: a Pilot RCT
Brief Title: ACT-DE for Diabetes Distress in Adults With Type 2 Diabetes: A Pilot RCT
Acronym: ACT-DE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anna Ngan, Principle Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACT-DE for Diabetes Distress
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Acceptance and Commitment Therapy; Type 2 Diabetes; Diabetes Distress
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants were random allocated (1:1 ratio) to either the intervention group that received a 6-week (5 sessions) group-based ACT-DE programme. While participants in the control group received 1 session of diabetes education.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor who is responsible for collecting outcome data and data entry has no idea about the group allocation of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT-DE (Experimental): The proposed intervention was a six-week acceptance-based diabetes education programme (ACT-DE) programme comprising Acceptance and Commitment Therapy (ACT) and diabetes education (DE). it included one diabetes education session (1st session), three ACT sessions (2nd to 4th), and a booster session in the 6th week conducted by the researcher. Each session lasted about 120 minutes in groups of 6 participants. The sessions were delivered face-to-face.
  Interventions: Behavioral: ACT-DE
- DE (Active Comparator): participants in the control group only received one session of diabetes education with the same session duration.
  Interventions: Behavioral: DE

INTERVENTIONS:
Behavioral: ACT-DE — The acceptance and commitment therapy is a psychological component to cultivate participants' acceptance attitude to diabetes and motivate them for a value-driven persistent diabetes self-management, directed by six psychological processes in the hexagonal model of ACT, including acceptance, cognitive defusion, the present moment, self-as-context, value clarification and committed action.
  Arms: ACT-DE
Behavioral: DE — DE
  Arms: DE

SUMMARY:
This study is a pilot RCT to examine the feasibility, acceptability and preliminary effectiveness of a 6-week acceptance-based diabetes education programme (ACT-DE) on diabetes distress, self-care efficacy and behaviours of adults with type 2 diabetes in Hong Kong.

It is hypothesise that the ACT-DE programme will:

* Be acceptable, feasible and beneficial for adults with type 2 diabetes to improve their psychological distress and self-care.
* Significantly reduce participants' diabetes distress (primary outcomes), when compared with the usual care (control) group immediately post-intervention;
* Significantly improve self-care efficacy, self-care behaviour and psychological flexibility (secondary outcomes) than the control group immediately post-intervention.

DETAILED DESCRIPTION:
Diabetes distress is an aversive feeling and emotional disturbance specific to diabetes, including the burden of daily self-care, worry and guilty feelings, and low satisfaction level with health care professionals. Around 36% of people with type 2 diabetes worldwide suffered from diabetes distress, which is associated with poor self-care performance, low self-efficacy in diabetes management and higher blood glucose levels. Acceptance and Commitment Therapy, one of the mindfulness and acceptance-based interventions, integrated with diabetes education are found to be potentially effective interventions for reducing diabetes distress.

Participants who agreed to participate in the study were randomly allocated into the intervention (N=24) and the control group (N=24). Participants in the intervention group received a 6-week group-based acceptance and commitment therapy integrated with diabetes education (ACT-DE). There were five sessions in 6 weeks with 120 minutes per session. The group size were 6. While participants in the control group received one session of diabetes education without any information on acceptance and commitment therapy.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling adults Hong Kong Chinese residents,
* aged 18-64,
* diagnosed with type 2 diabetes for over one year;
* at least moderate level of diabetes distress as measured with the Chinese Diabetes Distress Scale (CDDS-15; mean score >2 per item);
* having suboptimal blood glucose control as shown by HbA1c level of ≥ 7% in the laboratory results within the past six months;
* able to communicate in Cantonese and give written content.

Exclusion Criteria:

* history of a clinically diagnosed mental illness such as depression and anxiety disorder, and/or an acute/severe medical disease;
* noticeable cognitive impairment(s) as indicated by the total score (<6 of 10) of the Abbreviated Mental Test;
* recently received/receiving any psychological therapy such as mindfulness or acceptance-based therapy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female and Male
Enrollment: 48 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Diabetes Distress Scale | baseline (T0) and immediate post-intervention (T1)
  Diabetes distress was measured by the Chinese 15-item Diabetes Distress Scale (CDDS-15). It consists of 15 items rated on a six-point Likert scale from 1 = 'not a problem' to 6 = 'a serious problem'. A mean item score of 2-2.9 and ≥3.0 indicates moderate and severe distress, respectively.

SECONDARY OUTCOMES:
Diabetes self-management behaviours | baseline (T0) and immediate post-intervention (T1)
  was measured by the Chinese version of diabetes self-management activities (C-SDSCA). It has 11-items rated on an eight-point Likert scale from 0 to 7, with higher scores indicating more attention to self-management activities.
Diabetes management self-efficacy | baseline (T0) and immediate post intervention (T1)
  was measured by the Chinese version of Diabetes Management Self-Efficacy Scale (C-DMSES). The C-DMSES contains 20 items rated on an 11-point Likert scale, in which zero indicates not at all confident, and 10 indicates very confident.
Psychological flexibility | baseline (T0) and immediate post-intervention (T1)
  was measured by the Chinese version of the Acceptance and Action Questionnaire (AAQ-II Chinese). It contains seven items rated on a seven-point, agreement-based response scale from 1 = 'never true' to 7 = 'always true'. The AAQ-II will be scored by summing all item responses, with higher scale scores indicating a greater psychological inflexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Ms Anna Ngan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No